CLINICAL TRIAL: NCT04599153
Title: MRI-Volumetry in the Evaluation of Shunt Treatment for Hydrocephalus, a Randomised, Double-blind Study.
Brief Title: MRI-Volumetry in the Evaluation of Shunt Treatment for Hydrocephalus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Katarina Laurell, Senior Lecturer/Associate Professor, Uppsala University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Dnr 2017-254-31M
Record Dates: First submitted 2020-07-19; First posted 2020-10-22 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Hydrocephalus, Normal Pressure
Keywords: Ventriculoperitoneal Shunt; cerebral ventricular volume; cerebrospinal fluid
MeSH Terms: conditions — Hydrocephalus, Normal Pressure

STUDY DESIGN:
Intervention Model Description: Randomized, double blinded crossover design.
Who Masked: Participant, Outcomes Assessor
Masking Description: Shunt setting at the two months and three months follow up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High initial (Experimental): At the one month follow-up, the shunt is adjusted into a high opening pressure (2.5), which is crossed over to 1.0 at the two months follow-up. At the three months follow-up the opening pressure is set at 0.5 until the next day.
  Interventions: Other: Ventriculoperitoneal shunt opening pressure setting
- Low initial (Experimental): At the one month follow-up, the shunt is adjusted into a low opening pressure (1.0), which is crossed over to 2.5 at the two months follow-up. At the three months follow-up the opening pressure is set at 0.5 until the next day.
  Interventions: Other: Ventriculoperitoneal shunt opening pressure setting

INTERVENTIONS:
Other: Ventriculoperitoneal shunt opening pressure setting — The ventriculoperitoneal shunt (Strata®) opening pressure can be changed using a magnetic tool. The possible settings are 0.5, 1.0, 1.5, 2.0, 2.5 with a higher setting number corresponding to a higher opening pressure and less drainage through the shunt. All settings are used in routine clinical practice.

SUMMARY:
This randomized, double-blinded, cross-over study aim to evaluate the effects of shunt treatment in idiopathic normal pressure hydrocephalus (iNPH) by measuring cerebral ventricular volume and clinical symptoms at different shunt opening pressures. Further, proteins in the cerebrospinal fluid (CSF) will be compared before and after shunt surgery.

DETAILED DESCRIPTION:
The participants are evaluated before surgery and one month, two months, three months and three months plus one day after surgery. At each evaluation point a MRI of the brain with volumetric sequences is performed and clinical data is collected (Walking speed and steps for Time up and go, 10m walking and 3m walking backwards. Mini Mental State Examination, balance, gait, self rating of incontinence, Epworth Sleepiness Scale).

At surgery, all patients are given a ventriculoperitoneal (VP) shunt (Strata ® ) with an opening pressure setting of 1.5. After the first evaluation, one month postoperatively, participants are randomized to either a higher (2.5) or a lower (1.0) opening pressure, ratio 1:1. The opening pressure setting is blinded both for patients and the clinician during the subsequent clinical evaluations. At two months, the opening pressure is crossed over to the alternative setting (2.5 or 1.0). At three months, all participants receive the lowest shunt opening pressure (0.5) with the final evaluation the next day.

Semiautomatic measurement of the lateral as well as the third cerebral ventricles will be performed using the MRI scans and volumetric software: SyMRI (SyntheticMR AB, Linköping, Sweden)

CSF is collected at three times for each participant, from the lumbar spine pre- and 3 months postoperatively and intracranially during surgery. Further, intracranial CSF is taken through the Rickham Reservoir at the 3 months postoperative evaluation. After CSF from the participants has been collected, a single batch mass spectrometry will be performed with all the samples simultaneously.

Sample size was determined to achieve 80% power for a two tailed paired t-test for a mean change in ventricular volume of 8ml, estimated from postoperative change in ventricular volume in a previous study.

Hypotheses:

* The volume of the ventricular system in the brain decreases significantly after shunt-surgery.
* The ventricular volume is larger at high opening pressures compared to low opening pressures of the shunt.
* The decrease in ventricular volume is related to clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic normal pressure hydrocephalus and planned treatment with shunt surgery.

Exclusion Criteria:

* Ongoing anticoagulation treatment
* Ongoing Clopidogrel treatment
* Mini mental state examination results of 15 or lower.
* Contraindications to magnetic resonance imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-10-28 (Actual)

PRIMARY OUTCOMES:
Ventricular volume at different shunt settings (mL) | Assessed before surgery and at one, two and, three months and three months plus one day post surgery.
  Change in ventricular volume (ml) measured by MRI
Time of "Timed Up and Go" test at different shunt settings | Assessed before surgery and at one, two and, three months and three months plus one day post surgery.
  Change in total walking time (sec) on "Timed Up and Go".
Time of 10m walking test at different shunt settings | Assessed before surgery and at one, two and, three months and three months plus one day post surgery.
  Change in total walking time (sec) on 10m walking test.

SECONDARY OUTCOMES:
Ventricular versus lumbar cerebrospinal fluid composition determined by mass spectrometry | Cerebrospinal fluid is collected during diagnostic procedures before surgery, during surgery and three months and one day after surgery.
  Change in CSF composition from ventricular versus lumbar collection sites. Quantified with mass spectrometry and statistically compared on a protein by protein basis.
Change in CSF composition after surgery determined by mass spectrometry | Cerebrospinal fluid is collected during diagnostic procedures before surgery, during surgery and three months and one day after surgery.
  Change in CSF composition before versus after surgery. Quantified with mass spectrometry and statistically compared on a protein by protein basis.
Number of steps of "Timed Up and Go" test at different shunt settings | Assessed before surgery and at one, two and, three months and three months plus one day post surgery.
  Change in number of steps on "Timed Up and Go" test.
Number of steps of "Timed Up and Go" test at different time points regardless of shunt setting | Assessed before surgery and at one, two and, three months and three months plus one day post surgery.
  Change in number of steps on "Timed Up and Go" test.
Number of steps on 10m walking test at different shunt settings | Assessed before surgery and at one, two and, three months and three months plus one day post surgery.
  Change in number of steps on 10m walking test.
Number of steps on 10m walking test at different time points regardless of shunt setting | Assessed before surgery and at one, two and, three months and three months plus one day post surgery.
  Change in number of steps on 10m walking test.
Time of 3m backwards walking test at different shunt settings | Assessed before surgery and at one, two and, three months and three months plus one day post surgery.
  Change in total walking time (sec) on 3m backwards walking test.
Time of 3m backwards walking test at different time points regardless of shunt setting | Assessed before surgery and at one, two and, three months and three months plus one day post surgery.
  Change in total walking time (sec) on 3m backwards walking test.
Number of steps on 3m backwards walking test at different shunt settings | Assessed before surgery and at one, two and, three months and three months plus one day post surgery.
  Change in number of steps on 3m backwards walking test.
Number of steps on 3m backwards walking test at different time points regardless of shunt setting | Assessed before surgery and at one, two and, three months and three months plus one day post surgery.
  Change in number of steps on 3m backwards walking test.
Mini Mental State Examination at different shunt settings | Assessed before surgery and at one, two and, three months and three months plus one day post surgery.
  Change in Mini Mental State Examination results. (min 0, max 30, higher is better)
Mini Mental State Examination at different time points regardless of shunt setting | Assessed before surgery and at one, two and, three months and three months plus one day post surgery.
  Change in Mini Mental State Examination results. (min 0, max 30, higher is better)
Epworth sleepiness scale at different time points regardless of shunt setting | Assessed before surgery and at one, two and, three months and three months plus one day post surgery.
  Change in Epworth sleepiness scale rating. (min 0, max 24, lower is better)
Epworth sleepiness scale at different shunt settings | Assessed before surgery and at one, two and, three months and three months plus one day post surgery.
  Change in Epworth sleepiness scale rating. (min 0, max 24, lower is better)
Continence scale at different time points regardless of shunt setting | Assessed before surgery and at one, two and, three months and three months plus one day post surgery.
  Change in continence scale rating. (min 1, max 6, lower is better)
Continence scale at different shunt settings. | Assessed before surgery and at one, two and, three months and three months plus one day post surgery.
  Change in continence scale rating. (min 1, max 6, lower is better)
Balance scale at different shunt settings. | Assessed before surgery and at one, two and, three months and three months plus one day post surgery.
  Change in Balance scale rating. (min 1, max 7, lower is better)
Balance scale at different time points regardless of shunt setting | Assessed before surgery and at one, two and, three months and three months plus one day post surgery.
  Change in Balance scale rating. (min 1, max 7, lower is better)
Modified rankin scale at different time points regardless of shunt setting | Assessed before surgery and at one, two and, three months and three months plus one day post surgery.
  Change in Modified rankin scale rating. (min 0, max 6, lower is better)
Modified rankin scale at different shunt settings. | Assessed before surgery and at one, two and, three months and three months plus one day post surgery.
  Change in Modified rankin scale rating. (min 0, max 6, lower is better)
Gray matter volume at different time points regardless of shunt setting | Assessed before surgery and at one, two and, three months and three months plus one day post surgery.
  Change in whole brain grey matter volume measured by MRI (mL).
Gray matter volume at different shunt settings. | Assessed before surgery and at one, two and, three months and three months plus one day post surgery.
  Change in whole brain grey matter volume measured by MRI (mL).
White matter volume at different time points regardless of shunt setting | Assessed before surgery and at one, two and, three months and three months plus one day post surgery.
  Change in whole brain white matter volume measured by MRI (mL).
White matter volume at different shunt settings. | Assessed before surgery and at one, two and, three months and three months plus one day post surgery.
  Change in whole brain white matter volume measured by MRI (mL).
Time of "Timed Up and Go" test at different time points regardless of shunt setting | Assessed before surgery and at one, two and, three months and three months plus one day post surgery.
  Change in total walking time (sec) on "Timed Up and Go".
Time of 10m walking test at different time points regardless of shunt setting | Assessed before surgery and at one, two and, three months and three months plus one day post surgery.
  Change in total walking time (sec) on 10m walking test.
Ventricular volume at different time points regardless of shunt setting (mL) | Assessed before surgery and at one, two and, three months and three months plus one day post surgery.
  Change in ventricular volume (mL) measured by MRI

CONTACTS AND LOCATIONS:
Overall Officials: Katarina Laurell, MD, PhD, Principal Investigator — Uppsala University
Locations (1):
- Neurology Clinic, Östersund Hospital, Östersund, Jämtland County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liden S, Farahmand D, Laurell K. Volumetric effect of shunt adjustments in normal pressure hydrocephalus: a randomized, double-blind trial. J Neurosurg. 2023 Nov 17;140(5):1493-1500. doi: 10.3171/2023.9.JNS23668. Print 2024 May 1. PMID 37976516